CLINICAL TRIAL: NCT02294656
Title: Acute Pseudophakic Cystoid Macular Edema Treatment Trial: Intravitreal Ranibizumab Versus Triamcinolone Acetonide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Soll Eye (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML27905
Record Dates: First submitted 2014-11-04; First posted 2014-11-19 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: CYSTOID MACULAR EDEMA
Keywords: CYSTOID MACULAR EDEMA
MeSH Terms: conditions — Macular Edema | interventions — Ranibizumab; Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RANIBIZUMAB (Experimental): Ranibizumab patients will receive three monthly Ranibizumab 0.5 mg/0.05 mL injections, followed by PRN dosing, as treatment for acute pseudophakic cystoid macular edema.
  Interventions: Drug: Ranibizumab,
- TRIAMCINOLONE ACETONIDE (Active Comparator): Triamcinolone acetonide patients will receive PRN Triamcinolone acetonide 4 mg/0.1 mL injections, every 3 months, as treatment for acute pseudophakic cystoid macular edema.
  Interventions: Drug: Triamcinolone acetonide

INTERVENTIONS:
Drug: Ranibizumab, — Intravitreal injection of Ranibizumab as treatment for acute pseudophakic cystoid macular edema. Ranibizumab patients will receive three monthly Ranibizumab 0.5 mg/0.05 mL injections, followed by PRN dosing, as treatment for acute pseudophakic cystoid macular edema.
  Other Names: Lucentis
  Arms: RANIBIZUMAB
Drug: Triamcinolone acetonide — Intravitreal injection of Triamcinolone acetonide as treatment for acute pseudophakic cystoid macular edema. Triamcinolone acetonide patients will receive PRN Triamcinolone acetonide 4 mg/0.1 mL injections, every 3 months, as treatment for acute pseudophakic cystoid macular edema.
  Other Names: Triesence
  Arms: TRIAMCINOLONE ACETONIDE

SUMMARY:
This is an open-label, Phase I/II study evaluating intravitreal ranibizumab (R) vs. intravitreal Triesence (triamcinolone acetonide) (T) in subjects with acute pseudophakic cystoid macular edema (CME). Twenty consented patients with acute CME after phacoemulsification cataract surgery with posterior chamber intraocular lens implantation (PE/PCIOL) will be randomized 1:1 to treatment with R or T. R patients will receive three monthly R injections, followed by PRN dosing. T patients will receive PRN injections every 3 months. Clinical CME is defined as clinically evident CME, with visual acuity (VA) typically in the 20/40 to 20/200 range. Re-treatment criteria will include clinically evident worsening of CME, combined with any of the following:

* Any increase in spectral domain ocular coherence tomography (OCT) central macular thickness (CMT)
* Any observable fluid on OCT
* Any qualitatively increased perifoveal leakage/pooling on fluorescein angiography (FA).

Patients will be followed monthly through 12 months.

DETAILED DESCRIPTION:
1. BACKGROUND

   1.1 PATHOPHYSIOLOGY

   Despite improved cataract surgery instrumentation and techniques, the incidence of clinical CME remains 1 - 3% following uncomplicated PE/PCIOL. CME remains the most common cause of suboptimal post-operative visual acuity (VA) after uncomplicated PE/PCIOL. 1% clinical CME incidence represents 30,000 new cases annually in the USA. Clinical CME is defined as clinically evident CME, with VA typically 20/40 - 20/200. Diagnostic testing can confirm CME by FA leakage and increased CRT on OCT. If left untreated, chronic photoreceptor degeneration and irreversible VA loss can occur, even if the macular edema was to eventually resolve.

   1.2 TREATMENT OF PSEUDOPHAKIC CYSTOID MACULAR EDEMA Several treatment options for CME have been investigated, including topical, oral, periocular and intravitreal corticosteroids. Corticosteroids inhibit phospholipase A2, inhibiting production of arachidonic acid, precursor of the lipo-oxyenase (LOX) and cyclo-oxygenase (COX) pathways. Because corticosteroids inhibit both the LOX and COX pathways, corticosteroids may be expected to be more effective than non-steroidal anti-inflammatory drugs (NSAIDs) in decreasing inflammation. However, corticosteroids have side effects, including the potential for increased intraocular pressure (IOP) in susceptible patients, and require additional treatment for secondary glaucoma. NSAIDs specifically inhibit COX-2, and therefore avoid potential complications of corticosteroids. NSAIDs may be a good option for CME treatment of patients who are known corticosteroid responders. However, corneal stromal melting is a rare but serious potential side-effect of topical NSAIDs.

   1.3 RANIBIZUMAB (R) AND PSEUDOPHAKIC CYSTOID MACULAR EDEMA Numerous studies, such as ANCHOR, MARINA, and PIER, have shown that R effectively reduces perifoveal capillary leakage and CMT, when used as treatment for exudative age-related macular degeneration (AMD). BRAVO and CRUISE data have shown similar reduction in perifoveal capillary leakage and CMT when used as treatment for retinal vein occlusions (RVO).

   To date, there is no published study reporting efficacy of R monotherapy for acute pseudophakic CME. This study will assess R monotherapy, and eliminate any possible confounding effect of prior or concurrent treatment with either corticosteroids, NSAIDs, or both. Intravitreal R injections may avoid the potential for IOP elevation common with topical, periocular and intravitreal corticosteroids. R would also avoid corneal stromal melting, a rare but serious potential side-effect of topical NSAIDs.

   1.5 CLINICAL EXPERIENCE WITH RANIBIZUMAB R has been studied in more than 5000 subjects with neovascular AMD in a number of Phase I, I/II, II, III, and IIIb clinical trials. Serious adverse events related to the injection procedure have occurred in <0.1% of intravitreal injections, including endophthalmitis, rhegmatogenous retinal detachment (RD), and iatrogenic traumatic cataract. Other serious ocular adverse events observed among R-treated subjects and occurring in <2% of subjects include intraocular inflammation and increased IOP. The most common adverse reactions (reported > 6% higher in R-treated subjects than control subjects) were conjunctival hemorrhage, eye pain, vitreous floaters, increased IOP, and intraocular inflammation. Although there was a low rate (<4%) of arterial thromboembolic events (ATEs) observed in the R clinical trials, there is a potential risk of ATEs following intravitreal use of vascular endothelial growth factor (VEGF) inhibitors.
2. OBJECTIVES To assess the safety and efficacy of intravitreal ranibizumab (R) and triamcinolone acetonide (T) for treatment of acute pseudophakic CME.

   The primary objective of the study is to assess the SAFETY of intravitreal R and T for acute pseudophakic CME treatment, by evaluating:
   * Incidence and severity of ocular adverse events, as identified by eye examination
   * Incidence and severity of other adverse events, as identified by physical examination, subject reporting, and changes in vital signs

   The secondary objectives of the study are to determine EFFICACY of intravitreal R and T for acute pseudophakic CME treatment, by evaluating:
   * Mean change in spectral domain OCT CMT from baseline (microns)
   * Mean change in ETDRS letters from baseline (letters)
   * Proportion of patients with 3 line or better ETDRS letter improvement (%)
   * Time to 3 line ETDRS letter improvement (days)
   * Mean number of R or T injections (#)
   * Mean IOP (mm Hg)
3. STUDY DESIGN 3.1 DESCRIPTION OF THE STUDY This is an open-label, Phase I/II study evaluating intravitreal R vs. intravitreal T in subjects with acute pseudophakic CME. Twenty patients with acute CME after uneventful PE/PCIOL will be randomized 1:1 to treatment with R or T. R patients will receive three monthly R injections, followed by PRN dosing. T patients will receive PRN injections every 3 months.

   Re-treatment criteria will include clinically evident worsening of CME, combined with any of the following:
   * Any increase in spectral domain OCT CMT
   * Any observable fluid on OCT
   * Any qualitatively increased perifoveal leakage/pooling on FA. Patients will be followed monthly for 12 months.

   3.2 RATIONALE FOR STUDY DESIGN To date, there is no published study reporting efficacy of R monotherapy for acute pseudophakic CME. The proposed study would eliminate possible confounding effect of prior or concurrent treatment with steroids, NSAIDs, or both. Intravitreal R injections may avoid IOP elevation common with topical, periocular and intravitreal T injections.

   3.3 OUTCOME MEASURES

   3.3.1 Primary Outcome Measures

   The primary objective of the study is to assess the SAFETY of intravitreal R and T for acute pseudophakic CME treatment, by evaluating:
   * Incidence and severity of ocular adverse events, as identified by eye examination
   * Incidence and severity of other adverse events, as identified by physical examination, subject reporting, and changes in vital signs

   3.3.2 Secondary Outcome Measures

   The secondary objectives of the study are to determine EFFICACY of intravitreal R and T for acute pseudophakic CME treatment, by evaluating:
   * Mean change in spectral domain OCT CMT from baseline (microns)
   * Mean change in ETDRS letters from baseline (letters)
   * Proportion of patients with 3 line or better ETDRS letter improvement (%)
   * Time to 3 line ETDRS letter improvement (days)
   * Mean number of R or T injections (#)
   * Mean IOP (mm Hg)

   3.4 SAFETY PLAN All subjects will be queried as to systemic adverse events (AE). Potential ocular AE's predicted from common knowledge and historical data about R and T include: ocular injection, pain, discharge, redness, visual changes, floaters, IOP elevation, allergic reaction, infection, inflammation, RD, choroidal detachment, vitreous hemorrhage, and endophthalmitis. Potential systemic AE's include and are not limited to: stroke, heart attack, transient ischemic attack, reversible ischemic neurological defect, blood pressure elevation, weakness, headache, nausea, and malaise. AE incidence will be obtained by close examination and query of all subjects. All patients will be unmasked, so that any AEs will be readily apparent as to the causative drug. Testing and treatment recommendations will be made appropriate to the specific AE.

   3.5 COMPLIANCE WITH LAWS AND REGULATIONS This study will be conducted in accordance with current U.S. Food and Drug Administration (FDA) Good Clinical Practices (GCPs), and local ethical and legal requirements.
4. MATERIALS AND METHODS

4.1 SUBJECTS

4.1.1 Subject Selection 20 subjects from a single site will be enrolled. Eligible subjects will have been provided informed consent.

4.1.2 Inclusion Criteria

Subjects will be eligible if the following criteria are met:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Treatment naive subjects with a history of uncomplicated PE/CEIOL within 3 months of referral for treatment, and a diagnosis of CME secondary to PE/CEIOL within 1 month of referral for treatment.
* Best corrected VA 20/40 - 20/400.
* Spectral domain OCT CMT > 300 microns
* Treatment naive subjects with a history of uncomplicated cataract surgery within 12 months of referral for treatment and a diagnosis of CME secondary to cataract surgery within 12 months of referral for treatment.
* Patients who have received pre- or post-operative topical corticosteroids and/or NSAIDs will have to discontinue such medications for at least 2-4 weeks prior to entering this study.
* Best corrected ETDRS VA of 20/40 - 20/400.
* Spectral domain OCT central retinal thickness > 300 microns.

4.1.3 Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

* Diabetic retinopathy (DR) worse than moderate NPDR
* Macular edema associated with DR
* Ocular diseases causing decreased VA of the study eye, e.g. AMD or RD
* History of allergy to FA dye
* History of glaucoma surgery
* Active conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Concurrent use of systemic anti-VEGF agents
* Received any other experimental drug within 12 weeks prior to enrollment
* Currently being treated for active systemic infection
* Inability to comply with study or follow-up procedures
* Has a condition that, would preclude study participation (e.g. drug abuse)
* Pregnancy (positive pregnancy test) or lactation
* Pre-menopausal women not using adequate contraception
* Any condition that would pose a hazard to the subject if R or T were given
* Participation in another simultaneous medical trial

4.2 METHOD OF TREATMENT ASSIGNMENT

Patients will be randomized to treatment Group R or Group T according to the Treatment Randomization Chart in Appendix F:

* Group R: Three initial monthly injections followed by monthly PRN injections based on pre-defined retreatment criteria.
* Group T: One initial injection followed by PRN injections every 3 months based on pre-defined retreatment criteria.

All subjects will be unmasked to the treatment assignment.

4.3 STUDY TREATMENT

4.3.1 Formulation R is formulated as a sterile solution aseptically filled in a sterile, single use 2 mL stoppered glass vial. Each single use vial is designed to deliver 0.05 mL of 10 mg/mL ranibizumab aqueous solution with 10 mM histidine HCI, 10% trehalose dihydrate, and 0.01% polysorbate 20, pH 5.5.

T injectable suspension 40 mg/mL is a single use synthetic corticosteroid with anti-inflammatory action. Each mL of the sterile, aqueous suspension provides 40 mg of triamcinolone acetonide, with sodium chloride for isotonicity, 0.5% (w/v) carboxymethylcellulose sodium and 0.015% polysorbate 80. It also contains potassium chloride, calcium chloride (dihydrate), magnesium chloride (hexahydrate), sodium acetate (trihydrate), sodium citrate (dihydrate) and water for injection. Sodium hydroxide and hydrochloric acid may be present to adjust pH to a target value 6 - 7.5.

4.3.2 Dosage and Administration

a. Dosage Patients on R will receive 3 initial injections monthly followed by monthly PRN. Patients on T will receive an initial injection followed by PRN injections every 3 months.

Re-treatment criteria include clinically evident worsening of CME, combined with any of the following:

* Any increase in spectral domain OCT CMT
* Any observable fluid on OCT
* Any qualitatively increased perifoveal leakage/pooling on FA.

The intravitreal injection procedure will be carried out under controlled aseptic conditions. 0.5 mL of R will be given by intravitreal injection 3.0 to 3.5 mm posterior to the surgical limbus inferiorly. Similar technique will be used for T intravitreal injections, with two exceptions: one, a sterile 27-gauge ½ inch needle will be used for the intravitreal injection; and two, 4 mg T/0.1 mL volume will be injected intravitreally. Following the intravitreal injection, patients will be monitored for elevation in IOP and for endophthalmitis. Patients will be instructed to report any symptoms suggestive of endophthalmitis without delay.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible if the following criteria are met:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Treatment naive subjects with a history of uncomplicated cataract surgery within 3 months of referral for treatment and a diagnosis of CME secondary to cataract surgery within 1 month of referral for treatment.
* Best corrected ETDRS VA of 20/40 - 20/400.
* Spectral domain OCT central retinal thickness > 300 microns.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from this study:

* Any prior treatment for CME secondary to cataract surgery including but not limited to pre or post-operative corticosteroids, NSAIDS, etc.
* Subject has significant diabetic retinopathy (greater than moderate NPDR) or macular edema associated with diabetic retinopathy
* Any other additional ocular diseases which could irreversibly compromise the visual acuity of the study eye including anterior ischemic optic neuropathy (AION), age related macular degeneration (AMD), retinal detachment, etc.
* History of allergy to fluorescein, not amenable to treatment
* History of glaucoma surgery
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Concurrent use of systemic anti-VEGF agents
* Have received any other systemic experimental drug within 12 weeks prior to enrollment.
* Currently being treated for active systemic infection
* Inability to comply with study or follow-up procedures.
* Patient has a condition that, in the opinion of the investigator would preclude participation in the study (i.e. chronic alcoholism, drug abuse)
* Pregnancy (positive pregnancy test) or lactation
* Pre-menopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
SAFETY of INTRAVITREAL RANIBIZUMAB VS. TRIAMCINOLONE ACETONIDE FOR ACUTE PSEUDOPHAKIC CYSTOID MACULAR EDEMA TREATMENT (Incidence and severity of ocular adverse events) | 12 Months
  To assess the safety of intravitreal R and T for the treatment of acute pseudophakic cystoid macular edema by evaluating:
  * Incidence and severity of ocular adverse events, as identified by eye examination
  * Incidence and severity of other adverse events, as identified by physical examination, subject reporting, and changes in vital signs

SECONDARY OUTCOMES:
Mean change in spectral domain OCT CMT from baseline (microns) | 12 Months
  Mean change in spectral domain OCT CMT from baseline (microns)
Mean change in ETDRS letters from baseline (letters) | 12 Months
  Mean change in ETDRS letters from baseline (letters)
Proportion of patients with 3 line or better ETDRS letter improvement (%) | 12 Months
  Proportion of patients with 3 line or better ETDRS letter improvement (%)
Time to 3 line ETDRS letter improvement (days) | 12 Months
  Time to 3 line ETDRS letter improvement (days)
Mean number of R or T injections (#) | 12 Months
  Mean number of R or T injections (#)
Mean IOP (mm Hg) | 12 Months
  Mean IOP (mm Hg)

CONTACTS AND LOCATIONS:
Overall Officials: DAVID RHO, MD, Principal Investigator — Soll Eye
Locations (1):
- Soll Eye, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No